CLINICAL TRIAL: NCT06666088
Title: Program of Cognitive Stimulation and Strength Training on Cognitive Performance and Physical Mobility in Older Adults With Mild Cognitive Impairment
Brief Title: Cognitive Stimulation and Strength Training in Older Adults With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: -University Jaén.
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will not participate in the physical or cognitive exercise intervention but will receive general recommendations for comprehensive health care. This includes discussions about the benefits of engaging in physical and cognitive exercise, as well as advice on managing physical and mental health. All proposed physical and mental assessments will be conducted with the control group at the beginning of the study and after 12 weeks. Additionally, during the study period, they will be monitored for any changes in physical activity levels that may occur throughout the intervention. Follow-up will also include tracking nutritional changes, sleep habits, and stress levels.
- Experimental Group (Experimental): The experimental group will participate in a 12-week program combining cognitive stimulation and strength training, with two sessions per week. Each cognitive session, lasting 45 minutes to 1 hour, will aim to improve memory, attention, processing speed, and executive functions through activities like memory games and problem-solving tasks. A professional in neuropsychology or occupational therapy will lead these sessions, adapting activities to participants' abilities.
  Strength training will also be conducted twice a week for 45 minutes to 1 hour, focusing on exercises that strengthen major muscle groups and improve balance and coordination. Participants will use light weights, resistance bands, and bodyweight exercises, tailored to their physical levels. A specialized trainer will oversee the program, adjusting exercise intensity to ensure safety and optimize benefits.
  Interventions: Other: Cognitive stimulation and Strength training

INTERVENTIONS:
Other: Cognitive stimulation and Strength training — The experimental group will participate in a 12-week program to enhance cognitive functions and physical strength through twice-weekly sessions of 45 minutes to 1 hour. Cognitive stimulation activities will improve memory, attention, processing speed, and executive functions through memory games, recall exercises, and tasks that promote focus and quick thinking. Each session will be led by a neuropsychology or occupational therapy professional who will tailor activities to individual needs.
  Strength training will also occur twice a week, focusing on exercises that strengthen major muscle groups, improve balance, and enhance coordination. Participants will use light weights, resistance bands, and bodyweight exercises, with modifications based on their physical levels. A specialized trainer will supervise the program, progressively adjusting exercise intensity to ensure safety and optimize benefits.
  Arms: Experimental Group

SUMMARY:
This program focuses on integrating cognitive exercises and strength training for older adults experiencing mild cognitive impairment (MCI). It aims to enhance cognitive functions such as memory, attention, and problem-solving skills through various stimulating activities. At the same time, it incorporates strength training exercises to improve muscle mass, balance, and overall physical mobility. By addressing both cognitive and physical aspects of health, the initiative seeks to provide comprehensive benefits that may lead to improved quality of life for older adults with MCI. The research contributes valuable insights into the importance of holistic interventions in mitigating the effects of cognitive decline and promoting physical well-being in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* People over 60 years of age.
* Diagnosis of mild cognitive impairment (MCI) confirmed by neuropsychological evaluation or by a health professional.
* Ability to participate in moderate physical activities and perform strength exercises with supervision.
* Willingness and ability to regularly attend sessions of the cognitive stimulation and physical training program.
* Signed informed consent authorization, indicating that they understand and accept the objectives and activities of the program.

Exclusion Criteria:

* Diagnosis of moderate or severe dementia or other advanced cognitive impairment that prevents participation in the program.
* Severe or limiting physical conditions, such as heart disease, respiratory disease, or musculoskeletal injuries, that make it impossible to perform strength exercises.
* Psychiatric disorders (such as major depression or schizophrenia) or substance use that affect commitment or ability to follow the program activities.
* Participation in other cognitive stimulation or physical training programs or interventions in parallel, which may interfere with the evaluation of the effects of the program.
* Inability to understand and follow simple instructions, or lack of family or social support to attend the program if necessary.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Up to twelve weeks
  Instrument that examines the skills of attention, concentration, executive functions, memory, language, visuoconstructive abilities, calculation and orientation and the maximum score is 30.
Trail Making Test (TMT) | Up to twelve weeks
  It is used to assess executive function. It measures timed motor and visual tasks, and is divided into two tests: Part A (TMTA), which assesses speed and psychomotor attention and requires connecting consecutively numbered circles; and Part B (TMTB), which tests executive function and requires connecting alternating circles of numbers and letters. Longer completion times indicate poor performance.
Isaacs test | Up to twelve weeks
  Instrument used to assess verbal fluency. Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.Instrument used to assess verbal fluency. Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.
Mini-Mental State Examination (MMSE) | Up to twelve weeks
  The most widely used cognitive screening test to assess suspected symptoms consistent with cognitive impairment or dementia. Written test with a maximum score of 30. The cut-off point established for the MMSE defines "normal" cognitive function is generally set at 24, lower scores indicate more serious cognitive problems.
Tinetti Scale | Up to twelve weeks
  It is used to determine early the risk of falling in an elderly person during the year following its application. The result of both sections will be added, so that a score of less than 19 points will imply a high risk of falls, a score of 19 to 24 will reflect medium risk of falls and a score of 25 to 28 will indicate low risk of falls.
The Digit Symbol Substitution Test (DSST) | Up to twelve weeks
  Cognitive test to assess processing speed presented on a single sheet of paper that requires a subject to match symbols with numbers according to a key located at the top of the page. The subject copies the symbol into spaces below a row of numbers. The number of correct symbols within the allowed time, usually 90-120 seconds, constitutes the score.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess hand grip strength.
The Chair Stand Test (CST) | Up to twelve weeks
  It assesses leg strength, specifically the lower limb muscles, by evaluating a person's ability to repeatedly rise from a chair. The participant begins seated in a chair with their feet flat on the floor and their arms crossed over their chest. On command, they must stand up and sit down again as many times as possible in 30 seconds. The total number of repetitions completed is recorded as the test score. A higher number of repetitions indicates better lower limb strength. This test is commonly used to assess the functional capacity and balance of older adults, as leg strength is crucial for performing daily activities such as rising from a chair or walking.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Miguel Muñoz Perete, Jaén, Spain